CLINICAL TRIAL: NCT05741944
Title: The Value of a Risk Prediction Tool (PERSARC) for Effective Treatment Decisions of Soft-tissue Sarcomas Patients
Acronym: VALUE_PERSARC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, lvanbodegomvos, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL76563.058.21; 12642 (Other Grant/Funding Number: KWF Dutch Cancer Society); NL9160 (Registry Identifier: The Netherlands National Trial Register (NTR))
Record Dates: First submitted 2023-01-31; First posted 2023-02-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Soft-tissue Sarcoma; Predictive Cancer Model
MeSH Terms: conditions — Sarcoma | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care with the use of PERSARC (intervention) (Experimental): Patients in the intervention condition receive usual care with PERSARC added at two points in the decision making process. First, PERSARC will be used in multidisciplinary tumour boards (MTB) by STS professionals to guide treatment advice. Second, PERSARC will be used in patient consultations where the oncological/orthopaedic surgeon informs the patient about his/her diagnosis and discusses the benefits and harms of all relevant treatment options.
  Interventions: Other: Care with the use of PERSARC
- standard care (control) (Sham Comparator): All patients in the control condition receive standard care
  Interventions: Other: standard care

INTERVENTIONS:
Other: Care with the use of PERSARC — PERSARC is a personalized risk assessment tool which provides patients and STS professionals insight into the personalized risks and benefits of each treatment option based on patient's age, tumor size, tumor depth and histology. PERSARC will be used in multidisciplinary tumour boards to guide treatment advice and in consultation in which the oncological/orthopaedic surgeon informs the patient about his/her diagnoses and discusses the benefits and harms of all relevant treatment options
  Arms: Care with the use of PERSARC (intervention)
Other: standard care — All patients in control condition receive usual care.
  Arms: standard care (control)

SUMMARY:
The goal of this clinical trial is to assess the (cost-)effectiveness of a personalised risk assessment tool (PERSARC) to increase patients' knowledge about risks and benefits of treatment options and to reduce decisional conflict in comparison with usual care in high-grade extremity Soft-Tissue Sarcoma-patients.

High-grade (2-3) extremity Soft-Tissue Sarcoma patients (>= 18 years) will either receive standard care (control group) or care with the use of PERSARC; i.e. PERSARC will be used in multidisciplinary tumour boards to guide treatment advice and in consultation in which the oncological/orthopaedic surgeon informs the patient about his/her diagnoses and discusses the benefits and harms of all relevant treatment options (intervention group)

DETAILED DESCRIPTION:
To assess whether the use of the personalized risk assessment tool (PERSARC) is (cost)effective in reducing decisional conflict and increasing informed choices in high-grade extremity Soft-Tissue Sarcoma patients compared to usual care (co-primary outcomes). In addition, we aim to assess in a process evaluation (a) the involvement of patients in decision-making (b) the extent and way PERSARC is used by patients and professionals, and (c) how satisfied patients and professionals were with the use of PERSARC.

Study design: To assess the (cost)effectiveness of PERSARC in treatment decisions of high-grade extremity Soft-Tissue Sarcoma-patients, a parallel cluster randomized trial will be conducted in the 6 Dutch hospitals that are Soft-tissue sarcoma expertise centers. Hospitals will be randomized between standard care (control condition) or care with the use of PERSARC (intervention). Outcomes will be assessed within one week after treatment decision has been made (T1), and after 3, 6 and 12 months after the treatment decision has been made (T2, T3, T4) in at least 120 patients. See main study parameters/endpoints for a description of the outcomes that will be measured at these time points. Actual use of PERSARC, satisfaction with/added value of PERSARC and barriers and facilitators for the integration of PERSARC in treatment decision-making processes during patient-clinician encounters will be measured in a process evaluation using questionnaires, interviews, and audio-recording/observation of consultations.

Study population: Patients (>= 18 years) with primarily diagnosed (histologically confirmed) grade 2-3 extremity Soft-Tissue Sarcoma, who do not have a treatment plan yet and will be treated with curative intent. Patients with sarcoma subtypes or treatment options other than those mentioned in PERSARC are unable to participate. Furthermore, patients need to be Dutch fluency and literacy and mentally competent.

Intervention (if applicable): High-grade extremity Soft-Tissue Sarcoma patients will either receive standard care (control group) or care with the use of PERSARC; i.e. PERSARC will be used in multidisciplinary tumour boards to guide treatment advice and in consultation in which the oncological/orthopaedic surgeon informs the patient about his/her diagnoses and discusses the benefits and harms of all relevant treatment options (intervention group).

Main study parameters/endpoints: The co-primary outcomes are decisional conflict (Decisional Conflict Scale(DCS) (T1) and informed choice (T1). Informed choice is a combined outcome incorporating knowledge, attitudes concerning trade-offs between quality and length of life (QQ_Questionnaire) (T1), and treatment decision (T1). Secondary outcomes, include regret (Decision_Regret_Scale) (T3, T4), worry (Cancer_Worry_scale) (T1, T2, T3, T4), involvement in decision-making according to patients (SDM-Q-9) (T1), patient reported outcome using the Patient Reported Outcome Measures (PROMIS Global health) (T1, 2, 3, 4), and (PROMIS physical function) (T1, 2, 3, 4), utilities for the cost-effectiveness analysis (EQ-5D-5L) (T1, T2, T3, T4), health care cost (iMCQ) (T2, T3, T4) and absenteeism/presenteeism from paid work (T2, T3, T4).

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years
* Histologically diagnosed with grade 2-3 STS in their extremities.
* Who do not have a treatment plan yet
* Dutch fluency and literacy
* Mentally competent
* Signed informed consent
* Patient owns a phone with internet access (WiFi)

Exclusion Criteria:

* Patient that are treated without curative intent
* Patient that needs to be treated with chemotherapy or isolated limb perfusion
* Patients were surgery is not indicated
* Sarcoma subtypes not included in the PERSARC risk assessment tool

In summary: patients with sarcoma subtypes and/or patients that need to be treated with other treatment modalities than those included in the PERSARC risk assessment tool are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale | T1 (one week after treatment decision)
  Decisional conflict scale
  Items are given a score value of:
  strongly agree (0) - strongly disagree (4)
  Total score:
  16 items are a) summed, b) divided by 16, and c) multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict)
Informed choice | T1 (one week after treatment decision)
  combined outcome incorporating knowledge (self-developed questionnaire), attitudes concerning trade-offs between quality and length of life (QQ_Questionnaire, see below) and treatment decision
  self-developed knowledge questionnaire: a knowledge score was considered to reflect adequate decision-relevant knowledge if at least 50% of knowledge statements were correctly answered, which means a knowledge score ≥3 for the present study; no knowledge (0) - high knowledge (6)

SECONDARY OUTCOMES:
Decision Regret Scale | T3 (6m), T4 (12months)
  Decision Regret Scale
  Items are given a score value of:
  strongly disagree (1) - strongly agree(5)
  Total score:
  Scoring consist of reversing the scores of the 2 negatively phrased items, then taking the mean of the 5 items. These means were converted to a score ranging from 0 to 100 by subtracting 1 and multiplying by 25.
Cancer Worry Scale | T1 (one week after treatment decision), T2 (3months), T3 (6months), T4 (12months)
  Cancer Worry Scale
  Level of cancer worry was measured by the Dutch version of the Cancer Worry Scale, consisting of 6 questions with 4 response options (1 = not at all or rarely; 2 = sometimes; 3 = often; 4 = almost all the time), such that each individual attains a score ranging from 6 (minimum worry) to 24 (maximum worry).
SDM-Q-9 | T1 (one week after treatment decision), T2 (3months), T3 (6months), T4 (12months)
  Involvement in decision-making according to patients.
  Items are scored from completely disagree (0) to completely agree (5)
  Summing up all items leads to a raw total score between 0-45. Multiplication of the raw score by 20/9 provides a score forced (transformed) to range from 0 to 100, where 0 indicates the lowest possible level of SDM and 100 indicates the highest extent of SDM.
PROMIS Global health | T1 (one week after treatment decision), T2 (3months), T3 (6months), T4 (12months)
  Patient reported outcome measure
  10 item questionnaire lowest score (0) to highest (20). 0 Points represents the patient's most severe physical and/or mental impairment, while 20 represents the best possible state of health.
  The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores are indicative of a healthier patient.
PROMIS Physical function | T1 (one week after treatment decision), T2 (3months), T3 (6months), T4 (12months)
  Patient reported outcome measure
  10 item questionnaire lowest score (0) to highest (20).
  Scores are standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores are indicative of a healthier patient.
EQ-5D-5L | T1 (one week after treatment decision), T2 (3months), T3 (6months), T4 (12months)
  The EQ-5D-5L descriptive system comprises five dimensions (mobility, self-care, usual activities, pain and anxiety). Lowest score (1) - highest (5)
  Higher scores indicate unable to/ extreme problems
Medical consumption questionnaire (iMCQ) | T2 (3months), T3 (6months), T4 (12months)
  Medical consumption questionnaire (health care cost) focusing on healthcare use inside and outside the hospital. For the evaluation of cost, standard prices published in the Dutch costing guidelines will be used.
Productivity cost questionnaire (iPCQ) Cost of absenteeism from paid work will be calculated using the friction cost method. | T2 (3months), T3 (6months), T4 (12months)
  absenteeism/presenteeism from paid work

OTHER OUTCOMES:
process evaluation - a) the involvement of patients in decision-making | T1
  audio recordings of the patient-clinician consultation
  The audio-recordings of the patient consultations will be transcribed verbatim and assessed by two independent reviewers using the OPTION-5
process evaluation - b) the extent and way PERSARC is used by patients and professionals | end of study
  To gain insight into (b) the extent and way in which PERSARC is used by patients, user data from the VALUE-PERSARC app will be evaluated at group level (control vs intervention) (Google analytics within the app). Use of PERSARC by professionals will be examined through a checklist regarding the use of PERSARC in patient consultations and MTB
  Additionally, to gain further understanding of the integration of PERSARC in treatment decision making processes, 5-15 randomly selected patients and 3-4 STS professionals (one per intervention hospital) will be interviewed using a semi-structured interview scheme.
process evaluation - c) how satisfied patients and professionals were with the use of PERSARC | T1
  Satisfaction with the use of PERSARC (c) for patients and professionals who participated in the intervention arm and all professionals will be evaluated with a self-developed satisfaction questionnaire send to all eligible patients and professionals. Patients in the intervention arm will fill in the questionnaire within the VALUE-PERSARC app. Professionals are asked to fill in the questionnaire online, with reminders send after one week.

CONTACTS AND LOCATIONS:
Overall Officials: Leti van Bodegom-Vos, PhD, Principal Investigator — LUMC
Locations (7):
- Netherlands (7):
  - Radboud UMC, Nijmegen, Gelderland
  - Maastricht UMC, Maastricht, Limburg
  - Netherlands Cancer Institue, Amsterdam, North Holland
  - UMC Groningen, Groningen, Provincie Groningen
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of this trial, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provided a methodological sound proposal. Access needs to be requested at the Principal Investigator.

REFERENCES:
- [Derived] Kruiswijk AA, van de Sande MAJ, Haas RL, van den Akker-van Marle EM, Engelhardt EG, Marang-van de Mheen P, van Bodegom-Vos L; VALUE-PERSARC research group. (Cost-)effectiveness of an individualised risk prediction tool (PERSARC) on patient's knowledge and decisional conflict among soft-tissue sarcomas patients: protocol for a parallel cluster randomised trial (the VALUE-PERSARC study). BMJ Open. 2023 Nov 2;13(11):e074853. doi: 10.1136/bmjopen-2023-074853. PMID 37918933